CLINICAL TRIAL: NCT04107155
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effects of a Weight Management Program on Body Weight in Individuals Who Are Overweight and Otherwise Healthy
Brief Title: Study to Evaluate the Effects of a Weight Management Program on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CL100
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2019-09

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight | interventions — Suggestion; Diet, Healthy; Health Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Management Program (Experimental): Dietary Supplement: Saffron extract and Gynostemma extract with hesperidin and a handout with suggestions for healthy eating and overall health
  Interventions: Dietary Supplement: Weight Management Formulation; Other: Handout with Suggestions for Healthy Eating and Overall Health
- Placebo (Placebo Comparator): Placebo and handout with suggestions for healthy eating and overall health
  Interventions: Dietary Supplement: Placebo; Other: Handout with Suggestions for Healthy Eating and Overall Health

INTERVENTIONS:
Dietary Supplement: Weight Management Formulation — Saffron extract and Gynostemma extract with hesperidin
  Arms: Weight Management Program
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Other: Handout with Suggestions for Healthy Eating and Overall Health — Suggestions for Healthy Eating and Overall Health
  Arms: Weight Management Program
Other: Handout with Suggestions for Healthy Eating and Overall Health — Suggestions for Healthy Eating and Overall Health
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of the Weight Management Program on body weight

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled study to evaluate the effects of a Weight Management program on body weight. Each subject will receive a specific dose of the study product (A) to be taken twice daily with breakfast and dinner and a specific dose of the study product (B) to be taken 15 minutes before lunch daily for a total of 60 days. Each subject based upon the randomization will also receive a handout with suggestions for healthy eating and overall health.

Participants receive questionnaires, assessments, blood tests, vital signs and a body composition analysis.

The primary objective is the assessment of the change in body weight in response to the Weight Management program relative to baseline compared with placebo

The secondary objective is the assessment of the change in waist circumference, parameters from the body composition analysis, appetite, the levels of blood lipids and C-reactive protein in response to the Weight Management program relative to baseline compared with placebo

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, male or female, 21 - 70 years of age (volunteers between the ages of 71 and 75 inclusive will be permitted on a case-by-case basis at the discretion of the principal investigator).
2. A body mass index (BMI) of 25-34.9
3. Generally healthy and having no significant difficulty with digestion or absorption of food
4. Has been generally weight stable for the past six months (±6 lbs.)
5. Willing and able to give written informed consent
6. Clearly understands the procedures and study requirements
7. Willing and able to comply with all study procedures, including following the recommendations to maintain their usual diet and regular activity, as per protocol
8. Able to communicate, including reading, in English
9. Have not taken any nutritional supplements that may contain any of the components of the study product for a minimum of 14 days prior to baseline screening

Exclusion Criteria:

1. Having smoked any cigarette, electronic cigarette, cigar, pipe, or used a recreational drug or any product containing cannabidiol (CBD) or tetrahydrocannabinol (THC) in the past 30 days
2. Donation of blood within 30 days prior to screening/baseline
3. Inability to provide a venous blood sample
4. Participation in another study within 30 days prior to baseline/screening
5. Being pregnant or planning on becoming pregnant during study participation; or breast feeding
6. History of allergy or sensitivity to any component of the study products including saffron, dicalcium phosphate, gynostemma extract, hesperidin, microcrystalline cellulose, stearic acid, croscarmellose sodium, hydroxypropyl cellulose, vegetable cellulose, hypromellose, glycerin, silica, silicon dioxide, vegetable stearate, magnesium stearate or acacia gum
7. Currently taking a medication or dietary supplement specifically for weight loss and unwilling to washout (i.e. stop taking) for 14 days prior to baseline
8. Currently participating in a weight loss program and unwilling to discontinue participation prior to baseline
9. Having been diagnosed, received medical treatment or taking medication daily for the following medical condition(s):

   * Eating disorder (including anorexia nervosa, bulimia nervosa, binge eating disorder or avoidant or restrictive food intake disorder)
   * Psychiatric disorder
10. Presence of active or recurring clinically significant conditions as follows:

    * Diabetes mellitus or other endocrine disease
    * Eating disorder
    * Acute or chronic inflammatory disease or autoimmune disease
    * Cardiovascular disease including heart and blood vessel disease, arrhythmia, heart attack, stroke or heart valve problem
    * Gastrointestinal disease including gallbladder problems, gallstones or biliary tract obstruction
    * Thyroid disease (unless on a stable dose of medication for 3 months prior to screening and unlikely to change medication or dose during the study)
    * Hypertension (unless on a stable dose of medication for 3 months prior to screening and unlikely to change medication or dose during the study)
    * Neurologic condition/disease
    * Cancer (unless skin cancer other than melanoma which has been treated > 3 years prior to Baseline/screening)
    * Liver, pancreatic or kidney disease
    * Pulmonary disease
    * Blood coagulation disorder or other hematologic disease
    * Other condition or medication use that would preclude participation in the study in the judgment of the investigator/sub-investigator (Sub-I)
11. Currently taking any medications or treatment for a psychiatric disorder (bipolar disorder, manic disorder, schizophrenia, apathetic (inherited) disorder), that include antidepressant drugs, including the selective serotonin reuptake inhibitors (SSRIS), tricyclic and atypical antidepressants; benzodiazepines; central nervous system (CNS) depressants, dextromethorphan, meperidine, monoamine oxidase inhibitors (MAOIs); pentazocine, phenothiazines and tramadol. These may preclude participation in the study dependent on the judgment of the investigator/sub investigator.
12. Currently taking or having taken within the 30 days prior to screening/baseline any hormone replacement therapy (including dehydroepiandrosterone (DHEA), estrogen, progesterone, or testosterone; except those utilized as a method of birth control and which have been taken for > 3 months, with no anticipated change for the duration of the study)
13. Having had a surgical procedure or having an internal medical device which, in the judgment of the PI/Sub-I, would preclude participation in the study
14. Having abnormal screening laboratory test values including bilirubin > 2.5 x upper limit of normal (ULN), aspartate transaminase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine transaminase (ALT)/serum glutamic-pyruvic transaminase (SGPT) > 2.5 x ULN, serum creatinine > 1.5 mg/dL, blood glucose < 85 mg/dL or > 110 mg/dL, thyroid- stimulating hormone (TSH) level < 0.450 or > 4.500 milliunits per liter (mU/L) or other lab test result(s) that would preclude study participation in the judgement of the PI/Sub-I
15. Having blood pressure readings at Baseline/screening > 140 systolic or > 90 diastolic on two consecutive readings unless permitted to proceed to the next visit in the judgment of the PI/Sub-I
16. Currently consumes more than 7 standard alcoholic drinks per week for women and 14 drinks per week for men (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
17. Unable or unwilling to avoid consuming grapefruit juice or fresh grapefruit, Seville oranges and tangelos
18. History of known or suspected substance abuse (e.g. alcohol, opiates, benzodiazepines or amphetamines).
19. Having any other circumstance that precludes study participation in the judgment of the PI/Sub-I, including use of other nutritional supplements, which will be evaluated on a case-by-case basis.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Assessment of the mean change in Body Weight from baseline | 60 days
  Mean change from baseline to Day 60 in pounds from the Body Composition Analyzer

SECONDARY OUTCOMES:
Assessment of the mean change in Waist Circumference from baseline | 60 days
  Mean change from baseline to Day 60 in inches
Assessment of the mean change in Appetite from baseline | 60 days
  Mean change in the scores on a simplified nutritional appetite questionnaire from baseline. to Day 60. A numerical scale of 1-5 is used with the sum of the individual items totaling the score. A sum of less than or equal to 14 represents an improved score in support of weight loss.
Assessment of the mean change in the Total Cholesterol level from baseline | 60 days
  Mean change from baseline to Day 60 in mg/dL
Assessment of the mean change in the Triglyceride level from baseline | 60 days
  Mean change from baseline to Day 60 in mg/dL
Assessment of the mean change in the HDL Cholesterol level from baseline | 60 days
  Mean change from baseline to Day 60 in mg/dL
Assessment of the mean change in the LDL Cholesterol level from baseline | 60 days
  Mean change from baseline to Day 60 in mg/dL
Assessment of the mean change in the Total Cholesterol/HDL ratio from baseline | 60 days
  Mean change from baseline to Day 60 in ratio units
Assessment of the mean change in the Total Body Water from baseline | 60 days
  Mean change from baseline to Day 60 in pounds from the Body Composition Analyzer
Assessment of the mean change in the Lean Body Mass from baseline | 60 days
  Mean change from baseline to Day 60 in pounds from the Body Composition Analyzer
Assessment of the mean change in the Skeletal Muscle Mass from baseline | 60 days
  Mean change from baseline to Day 60 in pounds from the Body Composition Analyzer
Assessment of the mean change in the Body Fat Mass from baseline | 60 days
  Mean change from baseline to Day 60 in pounds from the Body Composition Analyzer
Assessment of the mean change in the Extracellular Water (ECW)/Total Body Water (TBW) ratio from baseline | 60 days
  Mean change from baseline to Day 60 in ratio units from the Body Composition Analyzer
Assessment of the mean change in the Basal Metabolic Rate from baseline | 60 days
  Mean change from baseline to Day 60 in kcal from the Body Composition Analyzer
Assessment of the mean change in the Visceral Fat Level from baseline | 60 days
  Mean change from baseline to Day 60 in the level from the Body Composition Analyzer
Assessment of the mean change in the Body Mass Index (BMI) from baseline | 60 days
  Mean change from baseline to Day 60 in (weight)kg/(height) m^2 from the Body Composition Analyzer
Assessment of the mean change in the Percent Body Fat from baseline | 60 days
  Mean change from baseline to Day 60 in the percent from the Body Composition Analyzer
Assessment of the mean change in the hs (high sensitivity)-C-reactive protein level from baseline | 60 days
  Mean change from baseline to Day 60 in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Swick, Ph.D, Principal Investigator — LIfe Extension
Locations (1):
- Life Extension Clinical Research, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aranganathan S, Nalini N. Efficacy of the potential chemopreventive agent, hesperetin (citrus flavanone), on 1,2-dimethylhydrazine induced colon carcinogenesis. Food Chem Toxicol. 2009 Oct;47(10):2594-600. doi: 10.1016/j.fct.2009.07.019. Epub 2009 Jul 24. PMID 19632289
- [Background] Carling D, Sanders MJ, Woods A. The regulation of AMP-activated protein kinase by upstream kinases. Int J Obes (Lond). 2008 Sep;32 Suppl 4:S55-9. doi: 10.1038/ijo.2008.124. PMID 18719600
- [Background] Chiranthanut N, Teekachunhatean S, Panthong A, Khonsung P, Kanjanapothi D, Lertprasertsuk N. Toxicity evaluation of standardized extract of Gynostemma pentaphyllum Makino. J Ethnopharmacol. 2013 Aug 26;149(1):228-34. doi: 10.1016/j.jep.2013.06.027. Epub 2013 Jun 21. PMID 23796877
- [Background] Dallal, G. (2017, July 10). www.Randomization.com. Retrieved from Randomization.com: http://www.randomization.com
- [Background] Ding, Y., Tang, K., Li, F., & et al. (2010). Effects of Gypenosides from Gynostemma pentaphyllum supplementation on exercise-induced fatigue in mice. African Journal of Agricultural Research, 5(6), 707-711.
- [Background] Diseases, N. I. (n.d.). www.niddk.nih.gov/health-information/weight-management. Retrieved May 6, 2019, from Weight Management: https://www.niddk.nih.gov/health-information/weight-management
- [Background] El-Marasy SA, Abdallah HM, El-Shenawy SM, El-Khatib AS, El-Shabrawy OA, Kenawy SA. Anti-depressant effect of hesperidin in diabetic rats. Can J Physiol Pharmacol. 2014 Nov;92(11):945-52. doi: 10.1139/cjpp-2014-0281. Epub 2014 Sep 19. PMID 25358020
- [Background] Food and Drug Administration. (2005, March 11). Guidance for Industry on Estimating the maximum safe starting dose in initial clinical trials for therapeutics in adult healthy volunteers. Federal Register, 70(140), 1-27. Retrieved from trc.
- [Background] Garg A, Garg S, Zaneveld LJ, Singla AK. Chemistry and pharmacology of the Citrus bioflavonoid hesperidin. Phytother Res. 2001 Dec;15(8):655-69. doi: 10.1002/ptr.1074. PMID 11746857
- [Background] Gauhar R, Hwang SL, Jeong SS, Kim JE, Song H, Park DC, Song KS, Kim TY, Oh WK, Huh TL. Heat-processed Gynostemma pentaphyllum extract improves obesity in ob/ob mice by activating AMP-activated protein kinase. Biotechnol Lett. 2012 Sep;34(9):1607-16. doi: 10.1007/s10529-012-0944-1. Epub 2012 May 11. PMID 22576281
- [Background] Ghasemi T, Abnous K, Vahdati F, Mehri S, Razavi BM, Hosseinzadeh H. Antidepressant Effect of Crocus sativus Aqueous Extract and its Effect on CREB, BDNF, and VGF Transcript and Protein Levels in Rat Hippocampus. Drug Res (Stuttg). 2015 Jul;65(7):337-43. doi: 10.1055/s-0034-1371876. Epub 2014 Apr 2. PMID 24696423
- [Background] Gout B, Bourges C, Paineau-Dubreuil S. Satiereal, a Crocus sativus L extract, reduces snacking and increases satiety in a randomized placebo-controlled study of mildly overweight, healthy women. Nutr Res. 2010 May;30(5):305-13. doi: 10.1016/j.nutres.2010.04.008. PMID 20579522
- [Background] Gynostemma Extract. (2015). Retrieved from UENSUN: http://naturalplantextract.com/herbal-extract/gynostemma-extract.html
- [Background] Hardie DG. AMP-activated protein kinase: a key system mediating metabolic responses to exercise. Med Sci Sports Exerc. 2004 Jan;36(1):28-34. doi: 10.1249/01.MSS.0000106171.38299.64. PMID 14707764
- [Background] Hardie DG. AMPK: a key regulator of energy balance in the single cell and the whole organism. Int J Obes (Lond). 2008 Sep;32 Suppl 4:S7-12. doi: 10.1038/ijo.2008.116. PMID 18719601
- [Background] Hardie DG. Sensing of energy and nutrients by AMP-activated protein kinase. Am J Clin Nutr. 2011 Apr;93(4):891S-6. doi: 10.3945/ajcn.110.001925. Epub 2011 Feb 16. PMID 21325438
- [Background] Hardie DG, Ross FA, Hawley SA. AMPK: a nutrient and energy sensor that maintains energy homeostasis. Nat Rev Mol Cell Biol. 2012 Mar 22;13(4):251-62. doi: 10.1038/nrm3311. PMID 22436748
- [Background] Hausenblas HA, Heekin K, Mutchie HL, Anton S. A systematic review of randomized controlled trials examining the effectiveness of saffron (Crocus sativus L.) on psychological and behavioral outcomes. J Integr Med. 2015 Jul;13(4):231-40. doi: 10.1016/S2095-4964(15)60176-5. PMID 26165367
- [Background] Hausenblas HA, Saha D, Dubyak PJ, Anton SD. Saffron (Crocus sativus L.) and major depressive disorder: a meta-analysis of randomized clinical trials. J Integr Med. 2013 Nov;11(6):377-83. doi: 10.3736/jintegrmed2013056. PMID 24299602
- [Background] Huyen VT, Phan DV, Thang P, Hoa NK, Ostenson CG. Antidiabetic effect of Gynostemma pentaphyllum tea in randomly assigned type 2 diabetic patients. Horm Metab Res. 2010 May;42(5):353-7. doi: 10.1055/s-0030-1248298. Epub 2010 Mar 8. PMID 20213586
- [Background] Imenshahidi M, Hosseinzadeh H, Javadpour Y. Hypotensive effect of aqueous saffron extract (Crocus sativus L.) and its constituents, safranal and crocin, in normotensive and hypertensive rats. Phytother Res. 2010 Jul;24(7):990-4. doi: 10.1002/ptr.3044. PMID 20013822
- [Background] Kaats GR, Miller H, Preuss HG, Stohs SJ. A 60day double-blind, placebo-controlled safety study involving Citrus aurantium (bitter orange) extract. Food Chem Toxicol. 2013 May;55:358-62. doi: 10.1016/j.fct.2013.01.013. Epub 2013 Jan 25. PMID 23354394
- [Background] Kamaraj S, Ramakrishnan G, Anandakumar P, Jagan S, Devaki T. Antioxidant and anticancer efficacy of hesperidin in benzo(a)pyrene induced lung carcinogenesis in mice. Invest New Drugs. 2009 Jun;27(3):214-22. doi: 10.1007/s10637-008-9159-7. Epub 2008 Aug 13. PMID 18704264
- [Background] Kianbakht, S., & Haiiaghaee, R. (2011). Anti-hyperglycemic effects of saffron and its active constituents, crocin and safranal, in alloxan-induced diabetic rats. Journal of Medicinal Plants, 3(39), 82-89.
- [Background] Kianbakht, S., & Mozaffari, K. (2009). Effects of saffron and its active constituents, crocin and safranal, on prevention of indomethacin-induced gastric ulcers in diabetic and nondiabetic rats. Journal of Medicinal Plants, 2(4), 30-38.
- [Background] Kola B. Role of AMP-activated protein kinase in the control of appetite. J Neuroendocrinol. 2008 Jul;20(7):942-51. doi: 10.1111/j.1365-2826.2008.01745.x. Epub 2008 Apr 28. PMID 18445126
- [Background] Lee WJ, Koh EH, Won JC, Kim MS, Park JY, Lee KU. Obesity: the role of hypothalamic AMP-activated protein kinase in body weight regulation. Int J Biochem Cell Biol. 2005 Nov;37(11):2254-9. doi: 10.1016/j.biocel.2005.06.019. PMID 16085448
- [Background] Li C, Schluesener H. Health-promoting effects of the citrus flavanone hesperidin. Crit Rev Food Sci Nutr. 2017 Feb 11;57(3):613-631. doi: 10.1080/10408398.2014.906382. PMID 25675136
- [Background] Li M, Lin XF, Lu J, Zhou BR, Luo D. Hesperidin ameliorates UV radiation-induced skin damage by abrogation of oxidative stress and inflammatory in HaCaT cells. J Photochem Photobiol B. 2016 Dec;165:240-245. doi: 10.1016/j.jphotobiol.2016.10.037. Epub 2016 Nov 1. PMID 27816646
- [Background] Li R, Li J, Cai L, Hu CM, Zhang L. Suppression of adjuvant arthritis by hesperidin in rats and its mechanisms. J Pharm Pharmacol. 2008 Feb;60(2):221-8. doi: 10.1211/jpp.60.2.0011. PMID 18237470
- [Background] Mashmoul M, Azlan A, Khaza'ai H, Yusof BN, Noor SM. Saffron: A Natural Potent Antioxidant as a Promising Anti-Obesity Drug. Antioxidants (Basel). 2013 Oct 29;2(4):293-308. doi: 10.3390/antiox2040293. PMID 26784466
- [Background] Mishra, R., Joshi, D., & Jiao, G. (2011). (Gynostemma pentaphyllum), The Chinese Rasayan-Current Research Scenario. International Journal of Research in Pharmaceutical and Biomedical Sciences, 2(4), 1483-1502.
- [Background] Miwa Y, Mitsuzumi H, Sunayama T, Yamada M, Okada K, Kubota M, Chaen H, Mishima Y, Kibata M. Glucosyl hesperidin lowers serum triglyceride level in hypertriglyceridemic subjects through the improvement of very low-density lipoprotein metabolic abnormality. J Nutr Sci Vitaminol (Tokyo). 2005 Dec;51(6):460-70. doi: 10.3177/jnsv.51.460. PMID 16521708
- [Background] Miwa Y, Yamada M, Sunayama T, Mitsuzumi H, Tsuzaki Y, Chaen H, Mishima Y, Kibata M. Effects of glucosyl hesperidin on serum lipids in hyperlipidemic subjects: preferential reduction in elevated serum triglyceride level. J Nutr Sci Vitaminol (Tokyo). 2004 Jun;50(3):211-8. doi: 10.3177/jnsv.50.211. PMID 15386934
- [Background] Lin-Na S, Yong-Xiu S. Effects of polysaccharides from Gynostemma pentaphyllum (Thunb.), Makino on physical fatigue. Afr J Tradit Complement Altern Med. 2014 Apr 3;11(3):112-7. doi: 10.4314/ajtcam.v11i3.17. eCollection 2014. PMID 25371572
- [Background] Nielsen IL, Chee WS, Poulsen L, Offord-Cavin E, Rasmussen SE, Frederiksen H, Enslen M, Barron D, Horcajada MN, Williamson G. Bioavailability is improved by enzymatic modification of the citrus flavonoid hesperidin in humans: a randomized, double-blind, crossover trial. J Nutr. 2006 Feb;136(2):404-8. doi: 10.1093/jn/136.2.404. PMID 16424119
- [Background] Ohara T, Muroyama K, Yamamoto Y, Murosaki S. Oral intake of a combination of glucosyl hesperidin and caffeine elicits an anti-obesity effect in healthy, moderately obese subjects: a randomized double-blind placebo-controlled trial. Nutr J. 2016 Jan 19;15:6. doi: 10.1186/s12937-016-0123-7. PMID 26786000
- [Background] Palit S, Kar S, Sharma G, Das PK. Hesperetin Induces Apoptosis in Breast Carcinoma by Triggering Accumulation of ROS and Activation of ASK1/JNK Pathway. J Cell Physiol. 2015 Aug;230(8):1729-39. doi: 10.1002/jcp.24818. PMID 25204891
- [Background] Park SH, Huh TL, Kim SY, Oh MR, Tirupathi Pichiah PB, Chae SW, Cha YS. Erratum: Antiobesity effect of Gynostemma pentaphyllum extract (actiponin): A randomized, double-blind, placebo-controlled trial. Obesity (Silver Spring). 2015 Dec;23(12):2520. doi: 10.1002/oby.21362. No abstract available. PMID 26727120
- [Background] Poirier P, Giles TD, Bray GA, Hong Y, Stern JS, Pi-Sunyer FX, Eckel RH; American Heart Association; Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Obesity and cardiovascular disease: pathophysiology, evaluation, and effect of weight loss: an update of the 1997 American Heart Association Scientific Statement on Obesity and Heart Disease from the Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2006 Feb 14;113(6):898-918. doi: 10.1161/CIRCULATIONAHA.106.171016. Epub 2005 Dec 27. PMID 16380542
- [Background] Razmovski-Naumovski, V., Hsun-Wei Huang, T., Tran, V., & et al. (2005). Chemistry and pharmacology of Gynostemma pentaphyllum. Phytochemistry Reviews, 4, 197-219.
- [Background] Rizza S, Muniyappa R, Iantorno M, Kim JA, Chen H, Pullikotil P, Senese N, Tesauro M, Lauro D, Cardillo C, Quon MJ. Citrus polyphenol hesperidin stimulates production of nitric oxide in endothelial cells while improving endothelial function and reducing inflammatory markers in patients with metabolic syndrome. J Clin Endocrinol Metab. 2011 May;96(5):E782-92. doi: 10.1210/jc.2010-2879. Epub 2011 Feb 23. PMID 21346065
- [Background] Rojas J, Arraiz N, Aguirre M, Velasco M, Bermudez V. AMPK as Target for Intervention in Childhood and Adolescent Obesity. J Obes. 2011;2011:252817. doi: 10.1155/2011/252817. Epub 2010 Dec 22. PMID 21318055
- [Background] Roohbakhsh A, Parhiz H, Soltani F, Rezaee R, Iranshahi M. Molecular mechanisms behind the biological effects of hesperidin and hesperetin for the prevention of cancer and cardiovascular diseases. Life Sci. 2015 Mar 1;124:64-74. doi: 10.1016/j.lfs.2014.12.030. Epub 2015 Jan 24. PMID 25625242
- [Background] Rosner, B. (n.d.). Hypothesis Testing: Two-Sample Inference-Estimation of Sample Size and Power for Comparing Two Means. In B. Rosner, Fundamentals of Biostatistics. Cengage Learning. Retrieved from www.stat.buc.ca: https://www.stat.ubc.ca/~rollin/stats/ssize/n2.html
- [Background] Shehata AS, Amer MG, Abd El-Haleem MR, Karam RA. The ability of hesperidin compared to that of insulin for preventing osteoporosis induced by type I diabetes in young male albino rats: A histological and biochemical study. Exp Toxicol Pathol. 2017 Apr 4;69(4):203-212. doi: 10.1016/j.etp.2017.01.008. Epub 2017 Jan 26. PMID 28132802
- [Background] Sheng L, Qian Z, Zheng S, Xi L. Mechanism of hypolipidemic effect of crocin in rats: crocin inhibits pancreatic lipase. Eur J Pharmacol. 2006 Aug 14;543(1-3):116-22. doi: 10.1016/j.ejphar.2006.05.038. Epub 2006 Jun 2. PMID 16828739
- [Background] Shirali S, Zahra Bathaie S, Nakhjavani M. Effect of crocin on the insulin resistance and lipid profile of streptozotocin-induced diabetic rats. Phytother Res. 2013 Jul;27(7):1042-7. doi: 10.1002/ptr.4836. Epub 2012 Sep 5. PMID 22948795
- [Background] U.S. Food & Drug Administration. (2018, April 1). CFR- Code of Federal Regulations Title 21. Retrieved from U.S. Department of Health and Human Services: https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/cfrsearch.cfm?cfrpart=182&showfr=1
- [Background] Ungvari Z, Parrado-Fernandez C, Csiszar A, de Cabo R. Mechanisms underlying caloric restriction and lifespan regulation: implications for vascular aging. Circ Res. 2008 Mar 14;102(5):519-28. doi: 10.1161/CIRCRESAHA.107.168369. PMID 18340017
- [Background] Visnagri A, Kandhare AD, Chakravarty S, Ghosh P, Bodhankar SL. Hesperidin, a flavanoglycone attenuates experimental diabetic neuropathy via modulation of cellular and biochemical marker to improve nerve functions. Pharm Biol. 2014 Jul;52(7):814-28. doi: 10.3109/13880209.2013.870584. Epub 2014 Feb 21. PMID 24559476
- [Background] Wang M, Wang F, Wang Y, Ma X, Zhao M, Zhao C. Metabonomics study of the therapeutic mechanism of Gynostemma pentaphyllum and atorvastatin for hyperlipidemia in rats. PLoS One. 2013 Nov 1;8(11):e78731. doi: 10.1371/journal.pone.0078731. eCollection 2013. PMID 24223845
- [Background] Xi L, Qian Z, Shen X, Wen N, Zhang Y. Crocetin prevents dexamethasone-induced insulin resistance in rats. Planta Med. 2005 Oct;71(10):917-22. doi: 10.1055/s-2005-871248. PMID 16254822